CLINICAL TRIAL: NCT01442129
Title: LVAD Therapy: Exploring the Effect of Intramyocardial Injection of Mesenchymal Precursor Cells on Myocardial Function
Brief Title: The Effect of Intramyocardial Injection of Mesenchymal Precursor Cells on Myocardial Function in Patients Undergoing LVAD Implantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deborah Ascheim (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Deborah Ascheim, Associate Professor, Clinical Director of Research, InCHOIR, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 08-1078-00006; U01HL088942 (NIH); U01HL088942-04 (NIH); 711 (Other: Ct Surgery Network Research Group)
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure; Cardiomyopathy; Ventricular Dysfunction
Keywords: Heart Failure; Left Ventricular Assist Device; Heart Transplantation; Cardiomyopathy; Destination Therapy; Cell Therapy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Ventricular Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPC Intramyocardial injection (Experimental): Intramyocardial injections of 25 million Mesenchymal Precursor Cells (MPCs)
  Interventions: Biological: MPC Intramyocardial injection
- Control Solution (Sham Comparator): Intramyocardial injections of 50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO
  Interventions: Biological: Control Solution

INTERVENTIONS:
Biological: MPC Intramyocardial injection — Intramyocardial injection of 25 million mesenchymal precursor cells at the time of LVAD implantation
  Other Names: RevascorTM
  Arms: MPC Intramyocardial injection
Biological: Control Solution — Injection of control solution during the LVAD implantation.
  Other Names: Cryoprotective media
  Arms: Control Solution

SUMMARY:
The main purpose of this research is to determine whether injecting mesenchymal precursor cells (MPC) into the heart during surgery to implant a left ventricular assist device (LVAD) is safe. MPCs are normally present in human bone marrow, and have been shown to increase the development of blood vessels and new heart muscle cells in the heart. In addition, this research is being done to test whether injecting the MPCs into the heart is effective in improving heart function.

DETAILED DESCRIPTION:
Intramyocardial injection of mesenchymal precursor cells (MPC) in patients with advanced heart failure who are treated with left ventricular assist device (LVAD) implantation may result in a renewable source of proliferating functional cardiomyocytes, as well as induce development of capillaries and larger size blood vessels to supply oxygen and nutrients to endogenous myocardium and newly-implanted cardiomyocytes, and release factors capable of paracrine signaling. If safety is established and an efficacy signal is observed in this exploratory trial, then the investigators will design a follow-up trial (stage 2) based on an adaptive design. The next trial would randomize patients to active therapy at one of two doses (25 and 75 million MPCs) versus placebo, and based on a predetermined selection criterion drop randomization to one of the dose arms as results accrue. Should this exploratory trial demonstrate safety but no signal of efficacy, then the subsequent trial would be based on a single dose of 75 million MPCs versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, inclusive of release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation;
* Age 18 years or older;
* If the subject or partner is of childbearing potential, he or she must be willing to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening and for a period of at least 16 weeks after procedure;
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening;
* Admitted to the clinical center at the time of randomization;
* Clinical indication and accepted candidate for implantation of an FDA approved implantable, non-pulsatile LVAD as a bridge to transplantation or for destination therapy.

Exclusion Criteria:

* Planned percutaneous LVAD implantation;
* Anticipated requirement for biventricular mechanical support;
* Cardiothoracic surgery within 30 days prior to randomization;
* Myocardial infarction within 30 days prior to randomization;
* Prior cardiac transplantation, LV reduction surgery, or cardiomyoplasty;
* Acute reversible cause of heart failure (e.g. myocarditis, profound hypothyroidism);
* Stroke within 30 days prior to randomization;
* Platelet count < 100,000/ul within 24 hours prior to randomization;
* Active systemic infection within 48 hours prior to randomization;
* Presence of >10% anti-human leukocyte antigen (anti-HLA) antibody titers with known specificity to the MPC donor HLA antigens;
* A known hypersensitivity to dimethyl sulfoxide (DMSO), murine, and/or bovine products;
* History of cancer prior to screening (excluding basal cell carcinoma);
* Acute or chronic infectious disease, including but not limited to human immunodeficiency virus (HIV);
* Received investigational intervention within 30 days prior to randomization;
* Treatment and/or an incompleted follow-up treatment of any investigational cell based therapy within 6 months prior to randomization;
* Active participation in other research therapy for cardiovascular repair/regeneration;
* Prior recipient of stem precursor cell therapy for cardiac repair;
* Pregnant or breastfeeding at time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, MD, Study Chair — Christiana Care Health Services; Patrick O'Gara, MD, Study Chair — Brigham and Women's Hospital
Locations (11):
- United States (11):
  - University of Florida, Gainsville, Florida
  - University of Maryland, Baltimore, Maryland
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Derived] Ascheim DD, Gelijns AC, Goldstein D, Moye LA, Smedira N, Lee S, Klodell CT, Szady A, Parides MK, Jeffries NO, Skerrett D, Taylor DA, Rame JE, Milano C, Rogers JG, Lynch J, Dewey T, Eichhorn E, Sun B, Feldman D, Simari R, O'Gara PT, Taddei-Peters WC, Miller MA, Naka Y, Bagiella E, Rose EA, Woo YJ. Mesenchymal precursor cells as adjunctive therapy in recipients of contemporary left ventricular assist devices. Circulation. 2014 Jun 3;129(22):2287-96. doi: 10.1161/CIRCULATIONAHA.113.007412. Epub 2014 Mar 28. PMID 24682346
- See also: Cardiothoracic Surgical Network Website — http://www.ctsurgerynet.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 11 U.S. centers with a Data and Clinical Coordinating Center (DCC); International Center for Health Outcomes and Innovation Research [InCHOIR], Icahn School of Medicine at Mount Sinai under an investigational new drug application. Enrollment began in May 2012, and the last patient was enrolled in August 2012.
Groups:
- MPC Intramyocardial Injection: Intramyocardial injections of 25 million MPCs
  Mesenchymal Precursor Cell Injection: Intramyocardial injection of 25 million mesenchymal precursor cells at the time of LVAD implantation
- Control Solution: Intramyocardial injections of 50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO
  50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO: Injection of control solution during the LVAD implantation.
Period: Overall Study
Arm/Group | MPC Intramyocardial Injection | Control Solution
Started | 20 | 10
Completed | 20 (Treatment withheld from 1 patient randomized before results of screening PRA known) | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with end-stage heart failure, either ischemic or non-ischemic etiology, who are being evaluated for LVAD implantation as a bridge-to-transplant (BTT) or destination therapy (DT)
Groups:
- Total: Total of all reporting groups
Arm/Group | MPC Intramyocardial Injection | Control Solution | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (15.4) | 62.2 (7.8) | 57.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 17 | 8 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
Cardiomyopathy [Number; unit: participants]
  Ischemic | 7 | 4 | 11
  Non-Ischemic | 13 | 6 | 19
Indication for LVAD [Number; unit: participants] — Bridge to Transplantation indicates that the LVAD is used to help patients in end stage heart failure who are awaiting a heart transplant.
  Destination Therapy indicates that the LVAD is planned for long-term use for patients in end stage heart failure who are not eligible for transplant.
  participants
    Bridge to Transplantation | 7 | 3 | 10
    Destination Therapy | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Intervention Related Adverse Events
Description: The primary safety endpoint of this study is the incidence of the following potential study-intervention related adverse events within 90 days post intervention (LVAD implantation + intramyocardial injection of study product): infectious myocarditis, myocardial rupture, neoplasm, hypersensitivity reaction, and immune sensitization.
Time Frame: 90 days
Measure: Number; unit: events
Arm/Group | MPC Intramyocardial Injection | Control Solution
Number analyzed (Participants) | 20 | 10
events | 0 | 0

2. Secondary Outcome: Functional Status and Ventricular Function
Description: The key efficacy endpoint of this study is functional status and ventricular function, while weaned from LVAD support, at 90 days post intervention (LVAD implantation + intramyocardial injection of study product). Functional status is defined by the ability to tolerate wean from LVAD support for 30 minutes without signs or symptoms of hypoperfusion, including, but not limited to symptoms of low output or signs of vascular congestion. Ventricular function will be assessed by transthoracic echocardiogram (TTE) in those patients able to be weaned for 30 minutes from LVAD support.
  The number of participants who successfully tolerated the 30 minute wean from LVAD support at 90 days is reported.
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | MPC Intramyocardial Injection | Control Solution
Number analyzed (Participants) | 20 | 10
participants | 10 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 months following randomization
Description: An independent Clinical Events Committee adjudicated adverse events and causes of death. Bleeding events were defined by transfusion of ≥ 4 units of packed cells within any 24 hour period during the first 7 days post LVAD implantation, and any transfusion of packed cells within any 24 hour period thereafter.
Arm/Group | MPC Intramyocardial Injection | Control Solution
Serious Adverse Events (participants affected / at risk) | 19/20 | 9/10
Other Adverse Events (participants affected / at risk) | 7/20 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPC Intramyocardial Injection (N=20) | Control Solution (N=10)
Major Bleeding (General disorders) | 8 (71) | 5 (30)
Cardiac Arrrest (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Fluid Collection (Cardiac disorders) | 3 (3) | 0 (0)
Device Malfunction - Pump Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hepatic Dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Major Infection - Localized Non-Device Infection (Infections and infestations) | 4 (4) | 2 (2)
Neurological Dysfunction - Other (Nervous system disorders) | 1 (1) | 0 (0)
Acute Renal Dysfunction (Renal and urinary disorders) | 4 (4) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Right Heart Failure (Cardiac disorders) | 3 (3) | 3 (3)
Venous Thromboembolism (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Baker's Cyst (General disorders) | 0 (0) | 1 (1)
Intraoperative Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Sustained Ventricular Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Sustained Supraventricular Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Device Malfunction - Non Pump Failure (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Device Malfunction - Pump Thrombus Suspected (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Device Malfunction - Pump Thrombus Confirmed (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Major Infection - Internal Pump Component Inflow or Outflow Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Major Infection (Infections and infestations) | 1 (1) | 0 (0)
TIA (Nervous system disorders) | 1 (1) | 0 (0)
Ischemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Toxic Metabolic Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Chronic Renal Dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0)
Elevated WBC, LDH (General disorders) | 1 (1) | 0 (0)
Shortness of Breath (General disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rib Pain (General disorders) | 1 (1) | 0 (0)
Sub-therapeutic Anticoagulation (General disorders) | 3 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPC Intramyocardial Injection (N=20) | Control Solution (N=10)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sustained Supraventricular Arrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hepatic Dysfunction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Localized Non-Device Infection (Infections and infestations) | 3 (5) | 2 (2)
Acute Renal Dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Venous Thromboembolism (Blood and lymphatic system disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No